CLINICAL TRIAL: NCT05723965
Title: Using CNN Image Recognition to Predict Rectal Cancer Outcomes
Brief Title: Using Artificial Intelligence to Predict Rectal Cancer Outcomes
Status: Completed | Type: Observational
Sponsor: Taichung Veterans General Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: CE21235B
Record Dates: First submitted 2023-01-05; First posted 2023-02-13 (Actual); Last update posted 2023-02-13 (Actual); Status verified 2023-02

CONDITIONS: Rectal Cancer Stage III
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- rectal cancer lesion images for training: Rectal cancer lesion images. Images with threatened (<2mm) circumferential margin of rectal cancer were labeled as "diseased". Otherwise, images were labeled as "normal". Using these materials as training materials for AI deep learning model buildup.
  Interventions: Other: As training material for deep learning model.
- rectal cancer lesion images for testing.: Using the buildup AI deep learning models from training cohort. Evaluating prediction rate of the model and analysis survival outcomes.
  Interventions: Other: As materials for external validation for the buildup model.

INTERVENTIONS:
Other: As training material for deep learning model. — Using labeled images as training materials for artificial intelligence to develop object detecting model.
  Groups: rectal cancer lesion images for training
Other: As materials for external validation for the buildup model. — Using the external validation set to evaluate prediction rate and survival outcome.
  Groups: rectal cancer lesion images for testing.

SUMMARY:
Investigator retrospective collect cases during 2010-2021 diagnosed as rectal adenocarcinoma with high quality CT images. Local advanced rectal cancer cases were labeled as "disease". Nor were defined " normal".

Using artificial intelligence CNN on jupyter notebook with open phyton code to train and develop models capable to recognizing local advanced rectal cancer. Modify the phyton code for better predict rate and help physician to quickly evaluate disease severity for fresh rectal cancer cases.

DETAILED DESCRIPTION:
From 2010.10.1~2021.12.31, rectal cancer patients with cT3-4 lesion was included. Collect high quality CT images with DICOM files in tumor segment. cT1-2, low rectal lesions, non-CRC cases were not included. Non-contrast and artificial defect images were also excluded. CT images were labeled as" diseased " when CRM were threatened (<2mm). All images were labeled according to judgment of 2 specialist. The data were separated into 2 parts. One for AI model training and testing, another for external validation. The training testing dataset was achieved by deep learning neural network and evaluating model accuracy performance. Then the model was applied into external validation dataset for real-world testing, evaluating coherent rate between AI and the Dr. decision. Furthermore, to see the cancer survival outcomes according to AI model prediction results.

ELIGIBILITY:
Inclusion Criteria:

* clinical staging T3-4 with high quality CT images.

Exclusion Criteria:

* 1. not primary malignancy lesion
* 2. not localizing rectum
* 3. T1-2 lesion
* 4. non contrast or poor quality images

Ages: 20 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Rectal cancer diagnosed during 2010.10.1-2022.7.31. clinical T3-4 lesion. with high quality CT images with contrast.
Sampling Method: Non-Probability Sample
Enrollment: 720 (Actual)
Dates: Start 2010-10-01 (Actual); Primary Completion 2022-07-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
accuracy of artificial intelligence with experienced physician | 1 week after images done.
  accuracy between artificial intelligence and experienced physician

SECONDARY OUTCOMES:
real life survival outcome of diagnosis by artificial intelligence. | 5 years after diagnosed
  real life survival outcome by artificial intelligence.

CONTACTS AND LOCATIONS:
Overall Officials: ChunuYu Lin, M.D., Principal Investigator — Taichung Veterans General Hospital
Locations (1):
- Taichung Verterans General Hospital, Taichung, Taiwan